CLINICAL TRIAL: NCT04919824
Title: Comparison of the Performance of Monopolar Current Cutting Knife and Bipolar RFA Knife in Colonic Endoscopic Submucosal Dissection
Brief Title: Monopolar Current Cutting Knife vs Bipolar RFA Knife
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mohamed Othman, MD, M.D. Director of Advanced Endoscopy Assistant Professor of Medicine - Gastroenterology Section, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-49483
Record Dates: First submitted 2021-05-20; First posted 2021-06-09 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Gastrointestinal Neoplasms
Keywords: Endoscopic Submucosal Dissection
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bipolar Knife (Experimental): ESD procedure performed with a novel bipolar knife.
  Interventions: Procedure: Endoscopic Submucosal Dissection; Procedure: Endoscopic Mucosal Resection
- Monopolar Knife (Active Comparator): ESD procedure performed with monopolar knives.
  Interventions: Procedure: Endoscopic Submucosal Dissection; Procedure: Endoscopic Mucosal Resection

INTERVENTIONS:
Procedure: Endoscopic Submucosal Dissection — Endoscopic submucosal dissection (ESD) is a novel technique for the removal of advanced colonic polyps with high-risk features. ESD is minimally invasive and allows the removal of colonic adenomatous polyp without resorting to surgery. The process of ESD includes marking the lesions selected for removal, followed by submucosal injection of a lifting agent, then circumferential incisions using a specialized knife followed by submucosal dissection of the entire lesion.
  Other Names: ESD
Procedure: Endoscopic Mucosal Resection — Endoscopic mucosal resection (EMR) is a conventional endoscopic technique commonly used for the resection of superficial neoplastic lesions in the GI tract. EMR carries lower morbidity and mortality compared to surgery.
  Other Names: EMR, Endoscopic resection

SUMMARY:
This is a prospective, randomized trial that aims to study the efficacy and clinical outcomes of a novel Bipolar Knife vs. Monopolar Knives on patients who undergo endoscopic submucosal dissection (ESD) procedure at Baylor St. Luke's Medical Center.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) is a novel technique for the removal of advanced colonic polyps with high-risk features. ESD is minimally invasive and allows the removal of colonic adenomatous polyp without resorting to surgery. The process of ESD includes marking the lesions selected for removal, followed by submucosal injection of a lifting agent, then circumferential incisions using a specialized knife followed by submucosal dissection of the entire lesion.

Traditionally, knifes utilizing monopolar current such as dual knife or hybrid knife were the preferred tools for endoscopic submucosal dissection. These knifes allows accurate dissection and excellent hemostasis. However, due to monopolar current generated heat, post coagulation syndrome can be seen in up to 8 to 40 % of patients. Post coagulation syndrome present with abdominal pain, fever and leukocytosis and requires supportive treatment with IV fluid and antibiotics. Recently, a novel bipolar Radiofrequency Ablation (RFA) knife were approved by FDA for the performance of ESD. The knife utilizes bipolar RFA current for submucosal dissection which can potentially expedite submucosal dissection and decrease the rates of post polypectomy syndrome.

Our tertiary referral center Baylor St Luke's Medical Center is center of excellence for ESD procedure and we have previously reported our ESD experience using specialized stability and traction device and monopolar current knife in 111 patients. The goal of our protocol is to compare the performance of monopolar current cutting knife and bipolar RFA knife in colonic endoscopic submucosal dissection.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years old
2. Patient is capable of providing informed consent
3. Patient is referred for ESD procedure of gastrointestinal neoplastic lesions

Exclusion Criteria:

1. Patient is < 18 years old
2. Patient refused and/or unable to provide consent
3. Patient is a pregnant woman
4. Patients with lesions removed with other techniques besides ESD or a modified ESD technique (i.e., EMR or TEM) as defined in the Japan Gastroenterological Endoscopy Society (JGES) guidelines for endoscopic resection of lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Procedure time | Day 1
  The speed of endoscopic submucosal dissection as calculated by cm2/hour

SECONDARY OUTCOMES:
Technical success rate | Day 1, 4 weeks
  En-bloc, R0 and curative resection rates for each knife
Procedural adverse event | Day 1
  Adverse events during the procedure: hemorrhage, perforation, etc.
Immediate post-procedural adverse event | Up to 24 hours
  Abdominal pain after the procedure using Visual Analogue Scale from 1 to 10
Delayed post-procedural adverse event | 4 weeks
  Post polypectomy syndrome in both groups up to one month after the procedure

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Baylor St. Lukes Medical Center (BSLMC), Houston, Texas

IPD SHARING:
Plan to Share IPD: No
This is a randomized prospective single-center study.

REFERENCES:
- [Background] Takeuchi Y, Uedo N, Ishihara R, Iishi H, Kizu T, Inoue T, Chatani R, Hanaoka N, Taniguchi T, Kawada N, Higashino K, Shimokawa T, Tatsuta M. Efficacy of an endo-knife with a water-jet function (Flushknife) for endoscopic submucosal dissection of superficial colorectal neoplasms. Am J Gastroenterol. 2010 Feb;105(2):314-22. doi: 10.1038/ajg.2009.547. Epub 2009 Sep 22. PMID 19773749
- [Background] Hong MJ, Kim JH, Lee SY, Sung IK, Park HS, Shim CS. Prevalence and clinical features of coagulation syndrome after endoscopic submucosal dissection for colorectal neoplasms. Dig Dis Sci. 2015 Jan;60(1):211-6. doi: 10.1007/s10620-014-3484-9. Epub 2014 Dec 13. PMID 25502119
- [Background] Jung D, Youn YH, Jahng J, Kim JH, Park H. Risk of electrocoagulation syndrome after endoscopic submucosal dissection in the colon and rectum. Endoscopy. 2013 Sep;45(9):714-7. doi: 10.1055/s-0033-1344555. Epub 2013 Aug 29. PMID 23990482
- [Background] Tsiamoulos ZP, Sebastian J, Bagla N, Hancock C, Saunders BP. A new approach to endoscopic submucosal tunneling dissection: the "Speedboat-RS2" device. Endoscopy. 2019 Jul;51(7):E185-E186. doi: 10.1055/a-0875-3352. Epub 2019 Apr 12. No abstract available. PMID 30978741
- [Background] Ismail MS, Bahdi F, Mercado MO, Habazi R, Alexander A, Prabhu S, John S, Kovvali C, Othman MO. ESD with double-balloon endoluminal intervention platform versus standard ESD for management of colon polyps. Endosc Int Open. 2020 Oct;8(10):E1273-E1279. doi: 10.1055/a-1226-6372. Epub 2020 Sep 22. PMID 33015328
- [Background] Cao Y, Liao C, Tan A, Gao Y, Mo Z, Gao F. Meta-analysis of endoscopic submucosal dissection versus endoscopic mucosal resection for tumors of the gastrointestinal tract. Endoscopy. 2009 Sep;41(9):751-7. doi: 10.1055/s-0029-1215053. Epub 2009 Aug 19. PMID 19693750
- [Background] Shinmura K, Ikematsu H, Kojima M, Nakamura H, Osera S, Yoda Y, Hori K, Oono Y, Ochiai A, Yano T. Safety of endoscopic procedures with monopolar versus bipolar instruments in an ex vivo porcine model. BMC Gastroenterol. 2020 Jan 31;20(1):27. doi: 10.1186/s12876-020-1176-9. PMID 32005163
- [Background] Williams CB, de Peyer RC. Bipolar snare polypectomy--a safer technique for electrocoagulation of large polyp stalks. Endoscopy. 1979 Feb;11(1):47-50. doi: 10.1055/s-0028-1098324. PMID 428352